CLINICAL TRIAL: NCT00438178
Title: A Phase I Study of Obatoclax Mesylate (GX15-070MS) in Patients With Acute Myeloid Leukemia (AML), Myelodysplastic Syndrome (MDS), Chronic Myeloid Leukemia (CML)in Myeloid Blast Phase, Myelofibrosis, Previously-Treated Chronic Lymphocytic Leukemia (CLL), or Aplastic Anemia
Brief Title: Safety and Efficacy of Obatoclax Mesylate (GX15-070MS) for the Treatment of Hematological Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gemin X (Industry)
Responsible Party: Jean Viallet, MD / Chief Medical Officer, Gemin X Pharmaceuticals
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GX006
Record Dates: First submitted 2007-02-21; First posted 2007-02-22 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Hematological Malignancies
MeSH Terms: conditions — Hematologic Neoplasms | interventions — obatoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Obatoclax mesylate (GX15-070MS)

SUMMARY:
Defects in the apoptotic process can lead to the onset of cancer by allowing cells to grow unchecked when an oncogneic signal is present. Obatoclax is designed to restore apoptosis through inhibition of the Bcl-2 family of proteins, thereby reinstating the natural process of cell death that is often inhibited in cancer cells.

DETAILED DESCRIPTION:
This is a multi-center, open-label, Phase I study of obatoclax administered every 2-week or weekly cycles, or as a Prolonged Infusion every 2 to 3 weeks to patients with Acute Myeloid Leukemia (AML), Myelodysplastic Syndrome (MDS), Chronic Myeloid Leukemia (CML)in Myeloid Blast Phase, Myelofibrosis, Previously-Treated Chronic Lymphocytic Leukemia (CLL), or Aplastic Anemia. Due to the PK/PD sampling schedule Cycle 1 will require overnight hospitalization. For the following cycles treatment may be administered on an outpatient basis but is at the discretion of the investigator. No investigational or commercial agents or therapies other than those described within the protocol may be administered with the intent to treat the patient's malignancy. Supportive care measures including those directed at controlling symptoms resulting from hematological malignancies are allowed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmation of AML, MDS, CML in blast phase, myelofibrosis, CLL, or aplastic anemia
* There are no limitations on additional, allowable type and amount of prior therapy as long as acute toxicities have resolved to the allowable grade.
* Must have normal organ functions
* Must be willing to submit to blood sampling for the planned PK and PD analyses.
* Must have the ability to understand and willingness to sign a written informed consent form

Exclusion Criteria:

* No other agents or therapies administered for the intent to treat
* Uncontrolled, intercurrent illness
* Pregnant women and women who are breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2005-10; Primary Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Determine the recommended Phase II dose of GX15-070MS; Characterize the DLTs of GX15-070MS; Determine the PK/PD response to GX15-070MS

SECONDARY OUTCOMES:
Describe any clinical responses of patient with hematological malignancies.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Viallet, MD, Study Director — Gemin X, Inc.
Locations (3):
- United States (2):
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - MD Anderson Cancer Center, Houston, Texas
- Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Result] Schimmer AD, O'Brien S, Kantarjian H, Brandwein J, Cheson BD, Minden MD, Yee K, Ravandi F, Giles F, Schuh A, Gupta V, Andreeff M, Koller C, Chang H, Kamel-Reid S, Berger M, Viallet J, Borthakur G. A phase I study of the pan bcl-2 family inhibitor obatoclax mesylate in patients with advanced hematologic malignancies. Clin Cancer Res. 2008 Dec 15;14(24):8295-301. doi: 10.1158/1078-0432.CCR-08-0999. PMID 19088047